CLINICAL TRIAL: NCT03509155
Title: A Multicenter Randomized Controlled Trial of Food Supplement Treatment for Wasting Children in Indonesia - Study Protocol
Brief Title: Food Supplement Treatment for Wasting Children in Indonesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SEAMEO Regional Centre for Food and Nutrition (Other)
Responsible Party: Principal Investigator, Muchtaruddin Mansyur, Principal Investigator, SEAMEO Regional Centre for Food and Nutrition
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PMT2017
Record Dates: First submitted 2018-03-12; First posted 2018-04-26 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Wasting; Nutrition Disorder, Child
Keywords: Infant and Young Child Feeding; Program Evaluation; Food Supplementation; Biscuit; wasting children
MeSH Terms: conditions — Cachexia; Child Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: The intervention is running parallel in three arms.
  1. The first arm as a control group obtaining only routine IYCF counseling by the cadre and without the provision of biscuits. If there are respondents at the first three months data collection who experience a decrease in nutritional status, then the respondent will be given biscuits immediately
  2. The second arm as the first intervention group to get biscuit with portion as recommended by Ministry of Health and also given the IYCF counseling by the cadres and nutritionist
  3. The third arm as the second intervention group receiving biscuit with adjustment in portion and IYCF Counseling that emphasize the optimization of local food In the 2nd and 3rd arm, treatment was administered for 3 months according to the recommended duration of biscuit delivery by the Ministry of Health, but all respondents from three arms will continue to be followed in third, sixth, and ninth months from the beginning of treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): The first arm as a control group obtaining only routine IYCF consultation by the posyandu (integrated health service post) cadres and without the provision of biscuits.
- National portion & IYCF counseling (Active Comparator): The second arm as the national portion & IYCF counseling group to get biscuit with standardized portion as recommended by Ministry of Health and also given the IYCF counseling by the cadres and nutritionist.In the second and third arm, treatment was administered for 3 months according to the recommended duration of biscuit delivery by the Ministry of Health, but all respondents from three arms will continue to be followed in third, sixth, and ninth months from the beginning of treatment.
  Interventions: Other: National portion & IYCF counseling
- Adjusted portion & local food counseling (Experimental): the third arm as the adjusted portion & local food counseling group receiving biscuit with adjustment in portion and IYCF Counseling that emphasize the optimization of local food. In the second and third arm, treatment was administered for 3 months according to the recommended duration of biscuit delivery by the Ministry of Health, but all respondents from three arms will continue to be followed in third, sixth, and ninth months from the beginning of treatment.
  Interventions: Other: Adjusted portion & local food counseling

INTERVENTIONS:
Other: National portion & IYCF counseling — Eight or twelve pieces of Biscuits supplementation per day as serving size recommendation based on the requirement from Ministry of Health, accompanied by IYCF Counseling emphasizing on local food optimization. The difference in serving size recommendation will be evaluated to see the efficacy of Biscuits supplementation on wasting children age 6-23 months of age
  Arms: National portion & IYCF counseling
Other: Adjusted portion & local food counseling — four pieces of Biscuits supplementation per day as serving size recommendation, accompanied by IYCF Counseling. The difference in serving size recommendation will be evaluated to see the efficacy of Biscuits supplementation on wasting children age 6-23 months of age
  Arms: Adjusted portion & local food counseling

SUMMARY:
Assessing program efficacy of under five food supplementation (PMT Biscuits) is needed after the first 6 months of exclusive breastfeeding, children were introduced to liquid and semi-solid food. In this phase of food introduction, children ability to accept food supplementation program was still questionable and the efficacy needs to be assessed.

Another aspect that needed to be evaluated is assessing the efficacy of food supplementation to improve the nutritional status of wasting children in multiple cities to describe Indonesian geographical and socio-economic diversity (multi center studies). PMT biscuits supplementation intervention is accompanied by educational modules on Infant and Young Child Feeding (IYCF) in order to improve caregiver's knowledge and skills in providing economically affordable and nutritious food for their children. PMT biscuits supplementation evaluation will be assessed at 9 months observations (3 months intervals). The observation will be conducted every month up until the first 3 months then the observation will be continued in 6th and 9th months of observation.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-17 months (still included in under two years old children during the intervention period)
* Underweight children by weight-per-height less than -2.00
* Not received PMT Biscuits at the time of recruitment
* Parents agree to follow the research

Exclusion Criteria:

* Severe wasting (weight for height less than -3 Z-score)
* Severe food insecurity households (Severe Household Food Insecurity)
* Tuberculosis infection based on anamnesis
* The possibility of moving to another city within 6 months of intervention

Ages: 6 Months to 23 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 720 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Nutritional status of wasting children | Through study completion, an average of 1 year. Measurement on changes in nutritional status from baseline and at third, sixth, & ninth months
  Anthropometry measurement based on weight-for-length indicator (The WHO Child Growth Standards). Weight will be measured in kilograms using an equivalent quality measurement tool using SECA scales. The measuring instrument to be used in measuring the length of the child is a Shorrboard with a unit of cm, precision of 0.1 cm.

SECONDARY OUTCOMES:
PMT biscuits compliance | Through study completion, an average of 1 year. At the first to third months after treatment started, then continued to be observed at the sixth and ninth months from the beginning of treatment.
  The caregiver will be asked to fill a form every day noting on how many biscuits the children eat and its remaining stock for that day. The form will be collected by enumerator while doing regular observation.

CONTACTS AND LOCATIONS:
Overall Officials: Muchtaruddin Mansyur, PhD, Principal Investigator — Seameo Regional Center For Food And Nutrition
Locations (1):
- Seameo Regional Center for Food and Nutrition, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de Onis M, Garza C, Victora CG. The WHO Multicentre Growth Reference Study: strategy for developing a new international growth reference. Forum Nutr. 2003;56:238-40. No abstract available. PMID 15806880
- [Background] Ferguson EL, Darmon N, Fahmida U, Fitriyanti S, Harper TB, Premachandra IM. Design of optimal food-based complementary feeding recommendations and identification of key "problem nutrients" using goal programming. J Nutr. 2006 Sep;136(9):2399-404. doi: 10.1093/jn/136.9.2399. PMID 16920861
- [Background] Fahmida U, Kolopaking R, Santika O, Sriani S, Umar J, Htet MK, Ferguson E. Effectiveness in improving knowledge, practices, and intakes of "key problem nutrients" of a complementary feeding intervention developed by using linear programming: experience in Lombok, Indonesia. Am J Clin Nutr. 2015 Mar;101(3):455-61. doi: 10.3945/ajcn.114.087775. Epub 2014 Dec 24. PMID 25733629
- [Background] Adu-Afarwuah S, Lartey A, Brown KH, Zlotkin S, Briend A, Dewey KG. Randomized comparison of 3 types of micronutrient supplements for home fortification of complementary foods in Ghana: effects on growth and motor development. Am J Clin Nutr. 2007 Aug;86(2):412-20. doi: 10.1093/ajcn/86.2.412. PMID 17684213
- [Derived] Kekalih A, Anak Agung Sagung IO, Fahmida U, Ermayani E, Mansyur M. A multicentre randomized controlled trial of food supplement intervention for wasting children in Indonesia-study protocol. BMC Public Health. 2019 Mar 13;19(1):305. doi: 10.1186/s12889-019-6608-5. PMID 30866888